CLINICAL TRIAL: NCT03212274
Title: A Phase 2 Study of the PARP Inhibitor Olaparib (AZD2281) in IDH1 and IDH2 Mutant Advanced Solid Tumors
Brief Title: Olaparib in Treating Patients With Advanced Glioma, Cholangiocarcinoma, or Solid Tumors With IDH1 or IDH2 Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01182; NCI-2017-01182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000023083; 10129 (Other: Yale University Cancer Center LAO); 10129 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Glioblastoma; Recurrent Cholangiocarcinoma; Recurrent Glioma; Recurrent Malignant Solid Neoplasm; WHO Grade 2 Glioma; WHO Grade 3 Glioma
MeSH Terms: conditions — Glioblastoma; Cholangiocarcinoma; Glioma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan and/or MRI, as well as a tumor biopsy and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo a MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib works in treating patients with glioma, cholangiocarcinoma, or solid tumors with IDH1 or IDH2 mutations that has spread from where it first started (primary site) to other places in the body (metastatic) and that does not respond to treatment (refractory). Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the overall response rates of olaparib in subjects with recurrent/progressive IDH1/2-mutant solid tumors, who will be recruited to 3 cohorts: a. glioma, b. cholangiocarcinoma, c. other solid malignant tumors.

SECONDARY OBJECTIVES:

I. To estimate the distribution of progression free survival (PFS) of olaparib in adults with recurrent/progressive IDH1/2-mutant glioma and cholangiocarcinoma.

II. To estimate the overall survival (OS) in adults with recurrent/progressive IDH1/2- mutant glioma and cholangiocarcinoma.

III. To determine the duration of response in adults with recurrent/progressive IDH1/2-mutant glioma, cholangiocarcinoma or other solid malignant tumors.

IV. To confirm the safety and tolerability of olaparib monotherapy.

EXPLORATORY OBJECTIVES:

I. To describe 2HG concentration in plasma by mass spectrometry at baseline and at specific timepoints and correlate with treatment response.

II. To describe 2HG levels in tumor biopsies from prior to the beginning of treatment and at specific timepoints and correlate with treatment response.

III. To evaluate in tumor biopsies and in liquid biopsies performed at baseline and at specific timepoints if co-occurring alterations detected via multiplexed immunofluorescence, mass cytometry (CyTOF)-imaging mass cytometry (IMC), ribonucleic acid (RNA) sequencing and/or deoxyribonucleic acid (DNA) sequencing can be associated with differential levels of 2HG production, treatment response and resistance.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a computer tomography (CT) scan and/or magnetic resonance imaging (MRI), as well as a tumor biopsy and blood sample collection on study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand the nature of this trial and provide written informed consent, prior to any study specific procedures; patients with Impaired Decision Making Capacity (IDMC) who have a close caregiver or legally authorized representative (LAR) may be considered eligible for this study at the treating physician's discretion, provided that the physician is reasonably sure that the possible risks and benefits of the study are clear and that the patient will take the drug as prescribed
* Subjects must be diagnosed with a glioma, cholangiocarcinoma or other solid malignant tumor that has progressed despite standard therapy, or for which no effective standard therapy exists, with biopsy-confirmed evidence of an IDH1 or IDH2 mutation associated with neomorphic activity of the encoded proteins; patients must have IDH1 or IDH2 mutation which must be detected in a clinical accredited laboratory using a Food and Drug Administration (FDA)-approved molecular test or a validated deoxyribonucleic acid (DNA)-based assay conducted in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory; only specific mutations that lead to a neomorphic phenotype will be eligible for enrollment, and include IDH1: R132V, R132G, R132S, R132L, R132C and R132H; IDH2: R140W, R140L, R140Q, R172W, R172G, R172S, R172M, R172K
* Patients must have tumors determined to be easily accessible for biopsy and must be willing to have serial biopsies (with a third biopsy upon evidence of disease progression); in case of multiple lesions, tumor biopsies will be performed on the most accessible site of disease; all possible precautions to avoid complications will be taken, including discussions in multidisciplinary meetings, if needed; patients affected by glioma will not be considered for study biopsies
* Patients must be willing to undergo extra blood sampling for correlative studies
* Subjects with extracranial disease must have evaluable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1); subjects affected by glioma must have evaluable disease by Response Assessment in Neuro-Oncology Criteria (RANO) criteria
* For subjects with glioma, specific inclusion criteria are as follows:

  * The disease should be recurrent or transformed glioma; subjects must not have had prior surgery (biopsy allowed) or radiation therapy within 3 weeks of enrollment
  * There must be an enhancing component of disease, as evaluated on pre-treatment magnetic resonance imaging (MRI)
  * For patients with World Health Organization (WHO) grade III or IV glioma and progressive disease < 12 weeks after completion of chemoradiotherapy, progression can be defined by the following set of criteria:

    * New enhancement outside of the radiation field (beyond the high-dose region or 80% isodose line)
    * If there is unequivocal evidence of viable tumor on histopathologic sampling (e.g., solid tumor areas. i.e., > 70% tumor cell nuclei in areas), high or progressive increase in MIB-1 proliferation index compared with prior biopsy, or evidence for histologic progression or increased anaplasia in tumor);
    * Note: Given the difficulty of differentiating true progression from pseudoprogression, clinical decline alone, in the absence of radiographic or histologic confirmation of progression, will not be sufficient for definition of progressive disease in the first 12 weeks after completion of concurrent chemoradiotherapy
  * For patients with WHO grade III or IV glioma and progressive disease >= 12 weeks after completion of chemoradiotherapy, progression can be defined by the following set of criteria:

    * New contrast-enhancing lesion outside of radiation field on decreasing, stable, or increasing doses of corticosteroids
    * Increase by >= 25% in the sum of the products of perpendicular diameters between the first post-radiotherapy scan, or a subsequent scan with smaller tumor size, and the scan at 12 weeks or later on stable or increasing doses of corticosteroids
    * For patients receiving antiangiogenic therapy, significant increase in T2/fluid attenuated inversion recovery (FLAIR) non-enhancing lesion may also be considered progressive disease; the increased T2/FLAIR must have occurred with the patient on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy and not be a result of comorbid events (e.g., effects of radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects)
    * Note: Clinical deterioration alone is not attributable to concurrent medication or comorbid conditions is sufficient to declare progression on current treatment but not for entry onto a clinical trial for recurrence
  * For patients with WHO grade II glioma progression is defined by any one of the following:

    * Development of new lesions or increase of enhancement (radiological evidence of malignant transformation)
    * A 25% increase of the T2 or FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not attributable to radiation effect or to comorbid events
* For subject with extracranial disease, they must have at least one lesion, not previously irradiated, that can be accurately measured at baseline as >= 10 mm in the longest diameter (except lymph nodes which must have short axis >= 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) or >= 10 mm with calipers by clinical exam OR at least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI/clinical exam at baseline and follow up visits
* Subjects must have progressive cancer at the time of study entry; prior experimental (non-FDA approved) therapies (other than drugs that share the same target) and immunotherapies are allowed; patients must not have received these therapies for 30 days or five half-lives of the drug (whichever is less) prior to the initiation of study treatment; toxicities from these therapies should have recovered to =< grade 1, with the exception of stable chronic grade 2 that is not overlapping with presumed toxicities of olaparib
* Female/male of age >= 18 years. This is because no dosing or adverse event data are currently available on the use of olaparib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) 0-2 (Karnofsky >= 50%)
* Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Leukocytes >= 3,000/mcL (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5 x ULN (within 28 days prior to administration of study treatment)
* Creatinine clearance estimated using the actual body weight and Cockcroft-Gault equation of >= 51 mL/min (within 28 days prior to administration of study treatment)
* Patients must have a life expectancy >= 16 weeks
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* No previous treatment with the specific assigned study drug or any other PARP inhibitor
* Prior radiation therapy is allowed; patients must not have received radiation therapy within 3 weeks prior to the initiation of study treatment
* Women of child-bearing potential are expected to use highly effective contraception during the study and for 1 month after the last dose of study drug; postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1; postmenopausal is defined as one or more of the following:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner

Exclusion Criteria:

* Patients should not enter the study if any of the following exclusion criteria are fulfilled
* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 30 days or five half-lives of the drug (whichever is less) prior to the initiation of study treatment (6 weeks for nitrosoureas or mitomycin C)
* Any previous treatment with PARP inhibitor, including olaparib
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for >= 5 years; patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Resting electrocardiogram (ECG) with corrected QT interval (QTc) > 470 msec or family history of long QT syndrome
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil); the required washout period prior to starting olaparib is 2 weeks; because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated drug information reference; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil); the required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents; because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated drug information reference; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Persistent toxicities caused by previous cancer therapy; toxicities should have recovered to =< grade 1, excluding alopecia and stable chronic grade 2 toxicity that is not overlapping with presumed toxicities of olaparib
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
* Patients with symptomatic uncontrolled brain metastases; a scan to confirm the absence of brain metastases is not required; the patient can receive a stable dose of corticosteroids before and during the study if these were started at least 4 weeks prior to treatment; patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days; patients with known uncontrolled brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Major surgery within 2 weeks of starting study treatment; effects from surgeries should have recovered to =< grade 1, with the exception of stable chronic grade 2 that is not overlapping with presumed toxicities of olaparib
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection; examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent and would limit compliance with study requirements
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Women who are actively breast feeding
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV); HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Olaparib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product; history of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib
* Patients with known active hepatitis (i.e. hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable)
* Patients who are receiving any other investigational agents
* Pregnant women are excluded from this study because olaparib is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib
* Patients with myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML), or features suggestive of MDS/AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to completion of course 8
  Will be determined by investigator assessment using Response Evaluation Criteria in Solid Tumors version 1.1 for extracranial solid tumors, Response Assessment in Neuro-Oncology criteria for intracranial glioma. Overall response rate and a 90% creditable interval in each cohort will be estimated using the approach described by Koyama. For the other solid tumors cohort, descriptive statistics and graphical displays will be used to summarize results within tumor types.

SECONDARY OUTCOMES:
Progression-free survival | From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  For time to event endpoints, Kaplan-Meier curves will be used to demonstrate distributions and median estimates will be reported with 95% confidence intervals. For each cohort, graphical displays such as swimmer plots, will be used to demonstrate patterns of response, progression and death, and in the third cohort they will also indicate disease type.
Incidence of adverse events | Up to 1 year
  Adverse events will be tabulated by type and grade in each cohort, and also across cohorts.

OTHER OUTCOMES:
2HG plasma magnetic resonance spectroscopy levels | Baseline up to post-treatment
  Absolute and fold changes for exploratory endpoints will be calculated between baseline and each subsequent follow-up time point. These will be displayed graphically versus (vs.) time for each cohort. Differences will be plotted vs. response status. Paired t-tests will be used to evaluate if differences between baseline and each subsequent time point are significant. Summary statistics will be reported (with 95% confidence intervals) to demonstrate mean differences in fold-change (or log fold-change) between responders and non-responders.
2HG plasma concentration level | Up to 1 year
  Absolute and fold changes for exploratory endpoints will be calculated between baseline and each subsequent follow-up time point. These will be displayed graphically vs. time for each cohort. Differences will be plotted vs. response status. Paired t-tests will be used to evaluate if differences between baseline and each subsequent time point are significant. Summary statistics will be reported (with 95% confidence intervals) to demonstrate mean differences in fold-change (or log fold-change) between responders and non-responders.
Co-occurring alterations | Baseline up to 1 year
  Will be detected via mass cytometry, ribonucleic acid sequencing and/or deoxyribonucleic acid sequencing. Will be associated with differential levels of 2HG production, treatment response and resistance. Absolute and fold changes for exploratory endpoints will be calculated between baseline and each subsequent follow-up time point. These will be displayed graphically vs. time for each cohort. Differences will be plotted vs. response status. Paired t-tests will be used to evaluate if differences between baseline and each subsequent time point are significant. Summary statistics will be reported (with 95% confidence intervals) to demonstrate mean differences in fold-change (or log fold-change) between responders and non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO
Locations (51):
- United States (51):
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin